CLINICAL TRIAL: NCT02165774
Title: Sacral Neuromodulation for Neurogenic Lower Urinary Tract Dysfunction: A Randomized, Placebo-controlled, Double-blind Clinical Trial
Brief Title: Sacral Neuromodulation for Neurogenic LUT Dysfunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: Insel Gruppe AG, University Hospital Bern (Other); Swiss Paraplegic Research, Nottwil (Network); Cantonal Hospital of St. Gallen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EK 2012 0048
Record Dates: First submitted 2014-06-02; First posted 2014-06-17 (Estimated); Last update posted 2018-01-09 (Actual); Status verified 2018-01

CONDITIONS: Refractory Neurogenic LUTD
Keywords: sacral neuromodulation, neurogenic lower urinary tract dysfunction

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- sacral neuromodulation ON (Active Comparator): active sacral neuromodulation (neuromodulator ON)
  Interventions: Device: Turning ON the neuromodulator
- sacral neuromodulation OFF (Placebo Comparator): placebo sacral neuromodulation (neuromodulator OFF)
  Interventions: Device: Turning OFF the neuromodulator

INTERVENTIONS:
Device: Turning OFF the neuromodulator — Turning OFF the neuromodulator in 50% of the patients in a randomized way by an investigator not involved in the assessment of the clinical outcome during the regular outpatient visit 2 months after neuromodulator implantation. It then follows a 2 months double-blind phase. Thereafter, i.e. during the regular outpatient visit 4 months after neuromodulator implantation, the unblinding takes place and in patients with sacral neuromodulation OFF, the neuromodulator is switched ON.
  Arms: sacral neuromodulation OFF
Device: Turning ON the neuromodulator
  Arms: sacral neuromodulation ON

SUMMARY:
Prospective, randomized, placebo-controlled, double-blind multicenter trial including 4 tertiary sacral neuromodulation referral centers in Switzerland (Zürich, Bern, Nottwil, St.Gallen). Patients with refractory neurogenic LUTD are included and randomized after neuromodulator implantation into sacral neuromodulation ON or sacral neuromodulation OFF (n=30) for a 2 months double-blind phase. In addition to standard neuro-urological assessments, patients who agree will also undergo neurophysiological investigation of the lower urinary tract, i.e. recording of current perception thresholds, sensory evoked potentials, and electroencephalography after stimulation of the urethra and bladder.

ELIGIBILITY:
Inclusion Criteria:

* Refractory neurogenic LUTD
* Urgency frequency syndrome and/or urgency incontinence refractory to antimuscarinics (pharmacotherapy for at least 4 weeks with at least 2 antimuscarinics)
* Chronic urinary retention refractory to alpha-blocker (pharmacotherapy with an alpha-blocker for at least 4 weeks)
* Combination of urgency frequency syndrome and/or urgency incontinence and chronic urinary retention refractory to antimuscarinics (pharmacotherapy for at least 4 weeks with at least 2 antimuscarinics) and alpha-blocker (pharmacotherapy with an alpha-blocker for at least 4 weeks)
* Stable neurological disease/injury for at least 12 months
* Age minimum 18 years
* Informed consent

Exclusion Criteria:

* Botulinum A toxin injections into the detrusor and/or urethral sphincter in the last 6 months
* Age under 18 years
* Pregnancy
* Individuals especially in need of protection (according to Research with Human Subjects published by the Swiss Academy of Medical Sciences)
* No informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2012-04; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Number of patients with successful sacral neuromodulation | 2 months
  success versus failure (yes/no variable)

CONTACTS AND LOCATIONS:
Locations (4):
- Switzerland (4):
  - Swiss Paraplegic Centre Nottwil, Nottwil, Canton of Lucerne
  - Cantonal Hospital of St. Gallen, Sankt Gallen, Canton of St. Gallen
  - University Hospital Inselspital Berne, Bern
  - University of Zurich, Balgrist University Hospital, Spinal Cord Injury Center, Zurich

REFERENCES:
- [Derived] Liechti MD, van der Lely S, Knupfer SC, Abt D, Kiss B, Leitner L, Mordasini L, Tornic J, Wollner J, Mehnert U, Bachmann LM, Burkhard FC, Engeler DS, Pannek J, Kessler TM. Sacral Neuromodulation for Neurogenic Lower Urinary Tract Dysfunction. NEJM Evid. 2022 Nov;1(11):EVIDoa2200071. doi: 10.1056/EVIDoa2200071. Epub 2022 Jul 7. PMID 38319849
- [Derived] Knupfer SC, Liechti MD, Mordasini L, Abt D, Engeler DS, Wollner J, Pannek J, Kiss B, Burkhard FC, Schneider MP, Miramontes E, Kessels AG, Bachmann LM, Kessler TM. Protocol for a randomized, placebo-controlled, double-blind clinical trial investigating sacral neuromodulation for neurogenic lower urinary tract dysfunction. BMC Urol. 2014 Aug 13;14:65. doi: 10.1186/1471-2490-14-65. PMID 25123172